CLINICAL TRIAL: NCT05925647
Title: The Effects of Mesenchymal Stem Cell Secretome in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, MD, Head of Hospital Research Unit, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAP06
Record Dates: First submitted 2023-03-09; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Messenchymal stem cell secretome
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: This study was divided into two groups, namely, control and treatment. Both received intervention in the form of a 1.5 cc injection on the scheduled day
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Mesenchymal stem cell placebo and secretome using injections that are similar in shape and color
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Messenchymal stem cell secretome (Experimental): The hypoxic mesenchymal stem cell secretome has been developed up to chapter 7, stored at -196 C to -135 C in cryopreservation, and has passed quality tests.
  Interventions: Drug: Messenchymal stem cell secretome
- Placebo (Placebo Comparator): Nacl 0,9% infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Messenchymal stem cell secretome — Mesenchymal stem cell secretome obtained from Kalbe Pharma Company
  Other Names: Messenchymal stem cell Concitioned Media
  Arms: Messenchymal stem cell secretome
Drug: Placebo — NaCl 0,9% infusion
  Other Names: NaCl 0,9% infusion
  Arms: Placebo

SUMMARY:
This research is a clinical trial of administering mesenchymal stem cell secretome to rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This research is experimental. The research subjects were 30 rheumatoid arthritis patients. The control group received a placebo, and the treatment group received mesenchymal stem cell secretome on the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 14th, 21st, and 28th. The data collected were erythroblastic acidity, hsCRP, interlukin 6, DAS-28, and assessment of drug side effects before and after therapy. Statistical test with paired difference test with p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis Patients

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Rheumatoid Arthritis Disease Activity | The change of Disease activity score patients at 1 months
  Disease Activity Score 28-joint count (DAS28) before and after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Moewardi General Hospital, Surakarta, Middle Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pratama YS, Pradiptakirana R, Rachmah A, Prabowo NA. Autoimmune Thrombocytopenia in SLE and COVID-19. Eur J Case Rep Intern Med. 2021 Nov 3;8(11):002863. doi: 10.12890/2021_002863. eCollection 2021. PMID 34912736
- [Result] Sholihah MM, Kusuma TRH, Hanif MI, Prabowo NA. Letter to the Editor on Type 1 diabetes onset triggered by COVID-19. Acta Diabetol. 2021 Sep;58(9):1283-1284. doi: 10.1007/s00592-021-01761-3. Epub 2021 Jun 28. No abstract available. PMID 34181079
- See also: Mesenchymal Stem Cell Conditioned Medium as Good as Methyl Prednisolone in Decreasing Levels of Interleukin 10 and The Degree of Pulmonary Vasculitis in Lupus Mice — https://www.banglajol.info/index.php/BJMS/article/view/51560